CLINICAL TRIAL: NCT05346055
Title: A Pilot Study of Delivering 'Engage' Psychotherapy Via Telemedicine Through the Tablet-based 'Prism' System to Homebound Older Adults With Depression
Brief Title: The Feasibility of Engage Therapy With Video Support for Homebound Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-10022828; 3P50MH113838-02S1 (NIH)
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Depression
Keywords: Older Adults
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Engage Prism 2.0 (Other): Engage Prism is a 9-week program that integrates Engage- a form of behavioral talk therapy treating depression, and guided use of Prism technology- a software that aims to improve social support and interaction of older adults.
  Interventions: Behavioral: Engage Prism (2.0)

INTERVENTIONS:
Behavioral: Engage Prism (2.0) — Brief Behavioral Treatment for Depression (Engage) combined with tablet-based social support system (Prism 2.0)

SUMMARY:
The primary aim in this pilot project is to test the feasibility, acceptability and impact (decreased depressive symptoms) of a brief behavioral treatment for depression (Engage) combined with video social support (PRISM 2.0) among socially isolated/lonely case management clients who endorse depressive symptoms. Eligible participants will be offered the combination of Engage and Prism 2.0, called Engage-Prism. The investigators hypothesize that the intervention (Engage Therapy With Video Support) will be accepted by participants, improve depressive symptom, and be feasible to complete.

DETAILED DESCRIPTION:
Engage is a brief therapy designed to offer a structured, stepped approach and interventions to reduce barriers to increased engagement with rewarding activities to improve depression (Alexopoulos et al, 2020). The goal is to increase participation in meaningful activities. Homebound older adults have limited social interaction given their restricted mobility and medical burden. In prior research with an intervention targeting social engagement with a technology intervention (PRISM 2.0), participants reported increased social support, decreased loneliness, increased feelings of well-being, more positive attitudes about computers, and gains in computer proficiency (Czaja et al., 2017).

Participants will be referrals from case management service. Clinicians will incorporate elements of the Prism system into therapy as appropriate, and participants will be instructed to use the Prism system at their leisure or as it pertains to their chosen "reward exposure" activities. There will be a post-therapy assessment and interview about their experience with the technology at week 9. The study will conclude with follow-up assessments at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 60 years
* English speaking
* Currently enrolled in case management at in 2 included agencies
* Major depression on the SCID
* 24-item Hamilton Depression Rating Scale (HAM-D) ≥ 19

Exclusion Criteria:

* Psychotic depression by SCID-V, i.e. presence of delusions
* High suicide risk, i.e. intent or plan to attempt suicide in the near future
* Presence of any Axis I psychiatric disorder
* Presence of substance abuse other than unipolar major depression
* History of psychiatric disorders, hypomania, are excluded
* Acute or severe medical illness, i.e. delirium, metastatic cancer, decompensated cardiac, liver, or kidney failure, major surgery, stroke, or myocardial infarction during the three months prior to entry; or drugs often causing depression, e.g. steroids, reserpine, alpha- methyl-dopa, tamoxiphen, vincristine
* Current involvement in psychotherapy
* Cognitive impairment (i.e. telephone administered MoCA < 11)
* Currently dwelling in non-community dwelling (e.g. prison, nursing home)
* Hearing that would not allow participants to complete sessions with the RA/therapist
* Vision impairment that would not allow the participant to use the study provided tablet
* Inability to speak English
* Aphasia interfering with communication
* Literacy -assessed by reading a paragraph designed for those at 6th grade reading level

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie C Benda, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results in publications after de-identification, as well as study protocol, treatment manuals, statistical analysis plan and informed consent.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After we publish the main results, we will make de-identified data available to other researchers under a data sharing agreement overseen by Weill Cornell Alacrity Center's executive committee.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. All researchers requesting data solely for research purpose; secure the data; return or destroy it once analyses are completed; do not share it with other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Virtual Senior Center, a community-building platform that helps older and homebound adults connect and engage with each other through virtual and hybrid classes. Recruitment efforts included online message board posts, emails, and virtual information sessions (via Zoom). Prospective participants contacted a study team member via phone or email and completed screening via phone. Participants were recruited between April 1, 2022 and June 30, 2022.
Period: Overall Study
Arm/Group | Engage Prism 2.0
Started | 8
Completed | 5
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Therapist decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Engage Prism 2.0
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.88 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7
  Black/African American | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Acceptability: Client Satisfaction Questionnaire (CSQ)
Description: The CSQ is a 3 - item questionnaire assessing client satisfaction with the treatment provided partway through the treatment (6 weeks). Scores range from 3 (least satisfied) to 12 (most satisfied).
Time Frame: 6 weeks (part-way through treatment)
Population: All participants completing the study were analyzed, although one participant is not included due to a database error. Those who did not complete the study could not complete the post-study CSQ.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage Prism 2.0
Number analyzed (Participants) | 4
score on a scale | 10.5 (4.34)

2. Primary Outcome: Acceptability: Client Satisfaction Questionnaire (CSQ)
Description: The CSQ is a 3 - item questionnaire assessing client satisfaction with the treatment provided assessed at 3 weeks post treatment (at 12 weeks) Scores range from 3 (least satisfied) to 12 (most satisfied).
Time Frame: 12 weeks (post treatment)
Population: Five total participants completed the study and 12-week follow up. Only 2 are included as three records were lost due to a databases error.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage Prism 2.0
Number analyzed (Participants) | 2
score on a scale | 9 (0)

3. Primary Outcome: Feasibility: Client Enrollment
Description: Feasibility will be measured as the number of clients who are referred to the program, meet eligibility and accept the intervention (versus refuse).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Engage Prism 2.0
Number analyzed (Participants) | 8
Participants | 8

4. Secondary Outcome: Hamilton Depression Rating Scale
Description: Change in depression scores from Baseline to 9 weeks. Scores range from 0 (no depression) to 54 (very severe depression).
Time Frame: Baseline, 9 weeks (end of treatment)
Population: Five participants completed this phase of the treatment, but only 3 are included as 2 were lost due to a database error.
Measure: Mean (Standard Deviation); unit: difference in pre/post score on a scale
Arm/Group | Engage Prism 2.0
Number analyzed (Participants) | 3
difference in pre/post score on a scale | 8.67 (2.52)

5. Secondary Outcome: Hamilton Depression Rating Scale
Description: Change in depression score from Baseline to 12 weeks post treatment. Scores range from 0 (no depression) to 54 (very severe depression).
Time Frame: Baseline, 12 weeks (post treatment)
Population: Five participants completed this phase of the treatment, but only 2 are included as 3 were lost due to a database error.
Measure: Mean (Standard Deviation); unit: difference in pre/post score on a scale
Arm/Group | Engage Prism 2.0
Number analyzed (Participants) | 2
difference in pre/post score on a scale | 0.5 (0.707)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the 9-week study period and 3-week follow up period (12 weeks total).
Arm/Group | Engage Prism 2.0
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT05346055/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT05346055/SAP_001.pdf